CLINICAL TRIAL: NCT05910905
Title: Evaluation of Clinical Efficacy of Preformed Pediatric Zirconia Crown and Preformed Pediatric Metal Crown: A Randomized Clinical Study
Brief Title: Clinical Efficacy of Preformed Pediatric Zirconia and Metal Crown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Haner Direskeneli, Professor, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17.05.23marmara
Record Dates: First submitted 2023-05-26; First posted 2023-06-20 (Actual); Last update posted 2023-06-20 (Actual); Status verified 2023-06

CONDITIONS: Carious Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prefabricated pediatric zirconia crown group (Experimental): Zirconia crowns (ZK; EZ Crowns, Spring Oral Health Technologies, Inc:, Loomis, Calif., USA).
  Interventions: Procedure: Prefabricated pediatric zirconia crown group
- Prefabricated stainless steel crown group (Active Comparator): Stainless Steel Crown (SSC, Kids Crown, Shinghung, Seoul, Korea)
  Interventions: Procedure: Prefabricated stainless steel crown group

INTERVENTIONS:
Procedure: Prefabricated pediatric zirconia crown group — Zirconia crown application: After preparing the molars, the crown was cemented by passive seating with modified glass ionomer cement (GC FujiCEM Evolve, GC America, Alsip, USA).
  Arms: Prefabricated pediatric zirconia crown group
Procedure: Prefabricated stainless steel crown group — Stainless steel crown application: After preparing the molars, the crown was filled with type-1 glass ionomer cement (Aqua Meron, Voco, Cuxhaven, Germany) and cemented.
  Arms: Prefabricated stainless steel crown group

SUMMARY:
The study was planned to evaluate and compare the clinical success of prefabricated stainless steel crowns and zirconia crowns used in the primary molars.

The study will be carried out in healthy children aged 6-9 years with caries on more than one surface of the primary molars.

DETAILED DESCRIPTION:
In this study, zirconia crowns will be compared with prefabricated stainless steel crowns in a randomized controlled manner. The study will be conducted in split-mouth to eliminate the effect of potential confounders. The obtained data will be analyzed using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 6-9 years with caries on primary molars
* Children without systemic disease or developmental dental anomalies that may affect caries susceptibility.
* Children whose cooperation is 'positive' or 'absolutely positive' according to the Frankl behavioral scale (Frankl et al., 1962).
* Those with deep dentin caries that do not extend to the pulp in the teeth to be treated
* The molars will be treated with a crown indication.
* Presence of symmetry of the primary molar to be treated in the opposite arch.
* The molar to be treated is in occlusion with the antagonist.
* Presence of caries on at least two surfaces of the molars to be treated.
* Absence of spontaneous pain, abscess, mobility, interradicular lesion in the tooth to be treated
* Patients whose parents and themselves agree to participate in the treatment

Exclusion Criteria:

* Children whose treatment cannot be continued on the dental chair due to cooperation
* Molars that will soon be exfoliated, 1/2 of the root has been resorbed
* The presence of bruxism
* The presence of erosion or attrition-related wear on the opposing molar
* The patient does not come to the control appointment or does not want to continue to the research
* Have allergy to local anesthetic, nickel or chromium
* Complications during treatment.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of clinical success | 24 month
  According to the criteria reported by Santamaria et al. (2004), clinical success will be categorized as successful, major failure, and minor failure.
  Successful:
  * No clinical signs or symptoms of pulp pathology
  * Tooth has exfoliated (without any minor/major failures)
  * No deformations in the crown/restoration
  * No pathology observed in radiographs
  Minor failure:
  * Reversible pulpitis (No need for root canal treatment or extraction)
  * Crown/restoration loss that can be restored
  * Presence of deformations/fractures/perforations in the crown/restoration
  * Permanent crown remaining submerged
  * Presence of new caries at the margins
  Major failure:
  * Irreversible pulpitis
  * Crown/restoration loss that cannot be restored
  * Inter-radicular radiolucency
  * Internal root resorption

SECONDARY OUTCOMES:
Parental satisfaction | 24 month
  To assess parental satisfaction regarding the applied restorations, scoring of crowns' appearance, color, shape, size, and general appearance will be requested using a Likert-type scale (Suguna & Gurunathan, 2021). Score 5 indicates the highest level of satisfaction, while score 1 represents the lowest level of satisfaction.
  1. Not at all satisfied
  2. Not satisfied
  3. Neither satisfied nor dissatisfied (Neutral)
  4. Satisfied
  5. Very satisfied

IPD SHARING:
Plan to Share IPD: No